CLINICAL TRIAL: NCT01839305
Title: Effects of Hydrotherapy on 3D Scapular Kinematics, Electromyography, Pain, Quality of Life, Balance and Cardiorespiratory Variables in Women With Fibromyalgia
Brief Title: Effects of Hydrotherapy on Physical Function and Quality of Life of Women With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mariana Arias Avila (Other)
Responsible Party: Sponsor-Investigator, Mariana Arias Avila, MSc, Universidade Federal de Sao Carlos
Organization: Universidade Federal de Sao Carlos (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 485/2011; FAPESP (Other Grant/Funding Number: 2011/22122-5)
Record Dates: First submitted 2013-04-17; First posted 2013-04-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Fibromyalgia
Keywords: Kinematics; Fibromyalgia; Physical Therapy; 3D Kinematics; Heart Rate Frequency; Hydrotherapy
MeSH Terms: conditions — Fibromyalgia | interventions — Hydrotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hidrotherapy (Experimental): Patients performed hydrotherapy 2 twice a week, for 16 weeks, to check if there was any effect on the outcome measures for women with fibromyalgia
  Interventions: Other: Hydrotherapy

INTERVENTIONS:
Other: Hydrotherapy — Hydrotherapy, monitored by physical therapists, performed in groups of up to 10 volunteers, for 45 min per session, twice a week, for 16 weeks

SUMMARY:
Fibromyalgia Syndrome (FS) is one condition that most affects functional performance, especially in women, due to alterations in the entire musculoskeletal system. Given that, Physical Therapy (PT) studies the human movement and its dysfunctions, and that FS, because of its complex chronic characteristic, impairs the affected individual's activities causing movement disorders, a PT professional must be part of the multidisciplinary team involved in the FS treatment. Nonetheless, as explained in the present proposal, several aspects still need clarification related to the PT role in this syndrome. Particularly, studies that analyze the biomechanical, sensorial and cardiorespiratory adaptations in individuals who undergo PT intervention still lack; those studies would contribute with scientific evidence to the clinical practice. According to recent systematic reviews, one of the most used therapies with positive effects on FS subjects is the hydrotherapy, which combines exercises and the water relaxing effects. Other alternative treatments have also been searched, in an attempt to decrease the painful picture presented, as the FS etiology and pathophysiology are not well known. The aim of this study is to evaluate the efficacy of different physical therapy resources in the FS, in two subprojects. The first will verify if hydrotherapy is effective in modifying movement variables (scapular kinematics and electromyography) and autonomic modulation. Other variables, such as pain level and quality of life in women with FS, will also be analyzed. The second study will evaluate the efficacy of the Shiatsu massage on pain, sleep quality, balance and quality of life of subjects with FS.

DETAILED DESCRIPTION:
Subjects were invited to take part in several assessments before starting the actual Hydrotherapy Treatment. These assessments were:

1. Three-dimensional scapular evaluation
2. Questionnaires (FIQ, SF-36, Beck Depression Inventory, Beck Anxiety Inventory, Pittsburgh Quality of Sleep Index)
3. Pain (pressure pain threshold and trigger points) Subjects were evaluated 3 times one month before starting treatment, one time in the middle of treatment and after treatment completion.

Treatment lasted 16 weeks and consisted of 2 weekly 45' hydrotherapy sessions.

ELIGIBILITY:
Inclusion Criteria:

* to have a clinical fibromyalgia diagnosis according to the 1990 ACR criteria
* to be aged from 30 to 60 years old.

Exclusion Criteria:

* Body Mass index >28kg/m²
* Cognitive deficits that prevented patients to understand the evaluation procedures
* Uncontrolled systemic illnesses (e.g. diabetes mellitus and systemic arterial hypertension)
* Neurological and musculoskeletal conditions that could have directly interfered in the evaluations, as paresis, important sensitive alterations, advanced joint diseases (e.g. arthroplasties or osteoarthritis)
* Infections
* Urinary incontinence
* Pregnancy

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2013-04 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Pain | up to 5 months from the initial interview
  Pain will be assessed as a composite measure through Visual Analogue Scale (VAS), Numerical Pain Rating Scale (NPRS), Myofascial Trigger Points (MTrPs) and Pressure Pain Threshold (PPT) on specific sites.

SECONDARY OUTCOMES:
3D Kinematics and electromyography | up to 5 months from the initial interview
  3D kinematics and electromyography will be evaluated with Flock of Birds, Motion Monitor Software and Delsys EMG Device

OTHER OUTCOMES:
Balance | up to 5 months from the initial interview
  Balance will be assessed by a force platform, in which patients will have to stand up still in some specific positions.
Function | up to 5 months from the initial interview
  Funtion will be assessed as a composite measure that includes questionnaires to evaluate different varibales that could be related to function: Fibromyalgia Impact Questionnaire, SF-36, Beck Depression Inventory, Beck Anxiety Inventory and Pittsburgh Sleep Quality Index.
Cardiorespiratory Status | up to 5 months from initial interview
  Cardiorespiratory status will be assessed by the heart rate variability, the ECG and the ergometric test

CONTACTS AND LOCATIONS:
Overall Officials: Tania F Salvini, PhD, Study Director — UFSCar; Antonio Roberto Zamunér, MSc, Principal Investigator — UFSCar; Deborah C Trevisan, MSc, Principal Investigator — UFSCar; Ester Silva, PhD, Study Chair — UFSCar; Paula R Camargo, PhD, Study Chair — UFSCar; Patricia Driusso, PhD, Study Chair — UFSCar
Locations (1):
- Academia O2, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zamuner AR, Andrade CP, Forti M, Marchi A, Milan J, Avila MA, Catai AM, Porta A, Silva E. Effects of a hydrotherapy programme on symbolic and complexity dynamics of heart rate variability and aerobic capacity in fibromyalgia patients. Clin Exp Rheumatol. 2015 Jan-Feb;33(1 Suppl 88):S73-81. Epub 2015 Mar 18. PMID 25786047